CLINICAL TRIAL: NCT04671810
Title: Prospective Observational Study of Long-term Pathogenic Treatment of Elizaria® in Patients With Paroxysmal Nocturnal Hemoglobinuria.
Brief Title: Prospective Observational Study of Long-term Pathogenic Treatment of Elizaria®
Acronym: NAP
Status: Completed | Type: Observational
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Other Study IDs: ECU-PNH-N01
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Elizaria® — Elizaria® will be prescribed by the Physician according to the actual SMPC.
  Other Names: Eculizumab

SUMMARY:
This is prospective observational study of long-term pathogenic treatment of Elizaria® in patients with paroxysmal nocturnal hemoglobinuria.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an ultra-rare, acquired, life-threatening, progressive clonal blood disease that is developed as a result of the expansion of one or more clones of hematopoietic stem cells with a somatic PIG A gene mutation. The main pathogenic mechanism of PNH development is a dysregulation of the complement system, in which there are no complement inhibitors CD55 and CD59 that are bounded by the GPI-anchor on the surface of blood cells, or there is a deficiency of them.

Eculizumab is the first drug for the pathogenetic therapy of PNH, a recombinant humanized monoclonal antibody against the C5 component of complement. Binding with high affinity to C5, eculizumab prevents the cleavage of C5 into C5a and C5b, thereby inhibiting the formation of pro-inflammatory cytokines (via C5a) and Membrane attack complex (MAC) (via C5b).

Using of eculizumab in patients with PNH leads to a significant decrease in hemolysis, the incidence of thrombosis and increasing of the quality of life of patients. It increases life expectancy with long-term using of eculizumab.

The drug Eculizumab, developed by JSC "GENERIUM", Russia, is a biological analogue (biosimilar) of the original drug Soliris®.

The population of the study is the patients with an established diagnosis of PNH who have indications for pathogenic treatment and are receiving Elizaria®.

The study duration for each patient will be at least 54 weeks for previously treated patients, and 58 weeks for previously untreated patients, including the Screening period and the observation period.

The study will include the Screening Period and the Observation Period:

* Screening Period - 2 weeks (Days 1 - 14);
* Follow-up is 52 weeks for previously treated patients and 56 weeks for previously untreated patients.

The screening period can be extended until the results of laboratory and instrumental studies are obtained, but no more than 14 days.

During the observation period, for the purpose of routine examination, it is planned to conduct a number of intermediate visits, approximately every 8 weeks (an acceptable interval of 6-10 weeks) between the Screening Visit (Visit 1) and the Study End Visit (Visit 13) in accordance with the plan of the dispensary observation of the patient. Additional visits and examinations may be carried out by the decision of the research physician.

If the patient is previously untreated, the patient undergoes induction therapy with Elizaria® at a dose of 600 mg weekly for 4 weeks with a further transition to maintenance therapy at a dose of 900 mg from the 5th week and then every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 2 years with an established diagnosis of PNH;
2. Prescribing Elizaria® as a pathogenetic therapy;
3. Signing by the patient of the informed consent form for participation in the study.

Exclusion Criteria:

1. Intolerance to eculizumab or other components of the drug.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of the study is the patients with an established diagnosis of PNH who have indications for pathogenic treatment and are receiving Elizaria®.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Dynamics of the peripheral blood LDH level during 52 weeks of the maintenance stage of treatment with Elizaria® (between Visits 6 and 13, inclusive). | 52-56 weeks
  To assess the dynamics of the peripheral blood LDH level during 52 weeks the area under the LDH level - time curve (AUC) will be calculated. Descriptive statistics will be provided for the values of the LDH level at each visit, as well as for the AUC, indicating the geometric means and coefficient of variation.

SECONDARY OUTCOMES:
Changes in hemoglobin levels during maintenance therapy with Elizaria® (between Visits 6 and 13 inclusive) | 52-56 weeks
  A paired t-test will be used to assess the change in hemoglobin level during the period of maintenance therapy with Elizaria® (between Visits 6 and 13, inclusive). Data on hemoglobin level and its change at each visit will be presented using descriptive statistics methods.
Number / proportion of patients with a change in the level of hemoglobin in the blood ± 5 g / l and ± 10 g / l. during the period of maintenance therapy with Elizaria® (between Visits 6 and 13 inclusive) | 52-56 weeks
  The proportion of patients with a change in blood hemoglobin level of ± 5 g / L and ± 10 g / L will be given during the period of maintenance therapy with Elizaria® (between Visits 6 and 13 inclusive).
The number / proportion of patients with various thrombotic complications that developed during treatment with Elizaria®. | 52-56 weeks
  For frequency indicators (the proportion of patients with various thrombotic complications) the absolute number of patients in the n / N format and the proportion of patients will be given and also calculated 95% confidence interval (CI) for the proportion.
The number / proportion of patients requiring transfusion of erythrocyte components of donated blood during treatment with Elizaria®. | 52-56 weeks
  For frequency indicators (the proportion of patients requiring transfusions of erythrocyte components of donated blood) the absolute number of patients in the n / N format and the proportion of patients will be given and also calculated 95% confidence interval (CI) for the proportion.
Number/proportion of patients with breakthrough hemolysis while observing an increased LDH, after a previous decrease in the course of treatment. | 52-56 weeks
  For frequency indicators (the proportion of patients with breakthrough hemolysis) the absolute number of patients in the n / N format and the proportion of patients will be given. and also calculated 95% confidence interval (CI) for the proportion.
Change in the size of PNH-clone of granulocytes and erythrocytes at Visits 6 and 13 relative to the initial value at screening. | 52-56 weeks
  To assess the dynamics of quantitative indicators (PNH-clone of granulocytes and erythrocytes, laboratory and vital indicators) relative to the initial level, a paired t-test or Wilcoxon's test will be used in case of a significant deviation from the normal distribution. The normal distribution will be tested using the Shapiro-Wilk test.
Frequency and severity of adverse events (AEs), serious adverse events (SAEs), including those associated with the use of Elizaria®, according to complaints, physical examination, assessment of vital signs, laboratory and instrumental studies, diaries. | 52-56 weeks
  Adverse events (AEs) that have developed since the patient signed the informed consent form will be coded using the MedDRA medical dictionary in the latest edition at the stage of database formation, until it is closed. The data on the incidence of AE / SAE during the course of the study will be presented by organ system (SOC) and preferred terms (PT) in terms of the number and proportion of patients who developed this adverse event. A summary of the severity of AEs and their relationship to treatment will be presented for each organ system.
Changes in vital signs, physical examination results, ECG, and laboratory values at Visit 13 from baseline at screening. | 52-56 weeks
  The number and proportion of patients with abnormalities according to complaints, physical examination, assessment of vital signs, laboratory and instrumental studies and patient diaries will be tabulated.
Number and proportion of patients with antidrug antibodies; titer of antidrug antibodies and their neutralizing activity. | 52-56 weeks
  For frequency indicators (the proportion of patients with antidrug antibodies) the absolute number of patients in the n / N format and the proportion of patients will be given and also calculated 95% confidence interval (CI) for the proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Markova, MD, Study Chair — AO GENERIUM
Locations (8):
- Russia (8):
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Chelyabinsk Oblast
  - State Budgetary Institution of Healthcare Irkutsk Order of the "Badge of Honor" Regional Clinical Hospital, Irkutsk, Irkutsk Oblast
  - State Budgetary Institution of Healthcare of the City of Moscow City Clinical Hospital named after S.P. Botkin of the Moscow Department of Health, Moscow, Moscow Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Novosibirsk State Medical University" of the Ministry of Health of the Russian Federation on the basis of the State Budgetary Institution of Health of the Novosibirsk Region "City Clinic, Novosibirsk, Novosibirsk Oblast
  - State budgetary institution of health care of the Republic of Karelia "Republican hospital named after V.A. Baranov ", Petrozavodsk, Republic of Karelia
  - State budgetary institution of the Rostov region "Rostov Regional Clinical Hospital", Rostov-on-Don, Rostov Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara, Samara Oblast
  - State Budgetary Healthcare Institution of the Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No. 1", Yekaterinburg, Sverdlovsk Oblast

IPD SHARING:
Plan to Share IPD: No